CLINICAL TRIAL: NCT00442039
Title: Pediatric Pharmacokinetic and Tolerability Study of Lithium for the Treatment of Pediatric Mania Followed by an Open Label Long Term Safety Period, Discontinuation Phase, and Restabilization Period.
Brief Title: Lithium for the Treatment of Pediatric Mania
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NICHD-2005-07-01; DUNS No. 07-775-8407
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Bipolar I Disorder Without Psychotic Symptoms
Keywords: Mania, Lithium, Bipolar, BPCA, pediatrics
MeSH Terms: conditions — Mania | interventions — Lithium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lithium dosing 1 (Experimental): The starting dose of lithium was 300 mg for patients weighing < 20 kg [no patients were enrolled that weighed less than 20 kg] and 600 mg for patients weighing ≥ 20 kg.
  Interventions: Drug: Lithium Carbonate
- Lithium dosing 2 (Experimental): The starting dose of lithium was 900 mg and the dose of lithium was increased weekly by 300 mg to maximum tolerated dose depending upon the patient"s response and tolerability.
  Interventions: Drug: Lithium Carbonate
- Lithium dosing 3 (Experimental): The starting dose of lithium was 900 mg and the lithium dose was increased by 300 mg every 3 days, (no more than twice weekly) to maximum tolerated dose based upon the patient"s response and tolerability.
  Interventions: Drug: Lithium Carbonate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lithium Carbonate — The starting dose of lithium was 300 mg for patients weighing < 20 kg
  Arms: Lithium dosing 1
Drug: Lithium Carbonate — The dose of lithium was increased weekly by 300 mg to maximum tolerated dose depending upon the patient"s response and tolerability. The starting dose of lithium was 900 mg and the dose of lithium was increased weekly by 300 mg to maximum tolerated dose depending upon the patient"s response and tolerability
  Arms: Lithium dosing 2
Drug: Lithium Carbonate — The starting dose of lithium was 900 mg and the lithium dose was increased by 300 mg every 3 days, (no more than twice weekly) to maximum tolerated dose based upon the patient"s response and tolerability.
  Arms: Lithium dosing 3
Drug: Placebo — During the third phase, which is the Discontinuation Phase, patients will be randomized to either placebo or lithium treatment for up to 28 weeks.
  Arms: Placebo

SUMMARY:
This clinical trial is being performed under the Best Pharmaceuticals for Children Act, signed into law in 2002 in order to improve pediatric labeling for off-patent drugs. The purpose of this study is to examine the efficacy and safety of lithium in the treatment of pediatric patients with bipolar I disorder.

DETAILED DESCRIPTION:
This is a multiphase, multicenter, trial that will comprehensively examine lithium in the treatment of pediatric patients with bipolar I disorder. In order to examine the treatment of bipolar disorder with lithium, this study will include four phases of treatment. The first phase, the Pharmacokinetic Phase, will include 8 weeks of Open Label treatment to determine empirically based dosing strategies for children and adolescents with bipolar disorder. Patients completing the Pharmacokinetic Phase, may be eligible to continue in the Long-Term Effectiveness Phase for a maximum of 16 weeks of lithium treatment. Subsequently, patients meeting response criteria during the Long-Term Effectiveness Phase will be eligible to continue in the Discontinuation Phase. During the Discontinuation Phase, patients will be randomized to either placebo or lithium treatment for up to 28 weeks. Finally, those subjects who experience a mood relapse during the Discontinuation Phase will be enrolled in an Open Label Restabilization Phase and treated with lithium for up to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. The patient was between the ages of 7 years and 17 years, 11 months at time of first dose.
2. The patient met DSM-IV diagnostic criteria, as assessed by a semi-structured assessment (Kiddie Schedule for Affective Disorders and Schizophrenia - Present and Lifetime [KSADS-PL]) and a separate clinical interview with a child/adolescent psychiatrist for manic or mixed episodes in Bipolar I disorder.
3. The patient had a score of ≥ 20 on the YMRS at screening and baseline.
4. The patient and legal guardian understood the nature of the study and were able to comply with protocol requirements. The legal guardian gave written informed consent and the youth, written assent.
5. Patients with comorbid conditions (attention deficit hyperactivity disorder [ADHD], conduct disorder) were eligible to participate.
6. If female: the patient was premenarchal, or was incapable of pregnancy because of a hysterectomy, tubal ligation, or spousal/partner sterility. If sexually active and capable of pregnancy, the patient must have been using an acceptable method of contraception (hormonal contraceptives, intrauterine device, spermicide and barrier) for at least 1 month prior to study entry and agreed to continue to use one of them for the duration of the study. If sexually abstinent and capable of pregnancy, the patient agreed to continue abstinence or to use of an acceptable method of birth control (either intrauterine device or spermicide and barrier) should sexual activity commence.
7. If female, the patient had a negative quantitative serum ß-human chorionic gonadotrophin hormone pregnancy test at screening and a negative qualitative urine pregnancy test at baseline, if female.
8. Patients with a history of substance abuse were eligible to participate if they agreed to continue to abstain from drugs during the trial and had a negative drug screen at screening or prior to baseline.
9. The patient was willing and clinically able to washout (approximately 5 half-lives) of exclusion medications during the screening period and prior to the administration of lithium. (No stable patients were asked to discontinue medications.)
10. The patient"s ECG and blood work (including complete blood count [CBC], electrolytes, etc.) showed no clinically significant abnormalities.

Exclusion Criteria:

1. The patient was clinically stable on current medication regiment for bipolar disorder.
2. The patient had a current or lifetime diagnosis of Schizophrenia or Schizoaffective Disorder, a Pervasive Developmental Disorder (Austin Screening Questionnaire score > 15), Anorexia Nervosa, Bulimia Nervosa, or Obsessive-Compulsive Disorder.
3. The patient had a current DSM-IV diagnosis of Substance Dependence.
4. The patient had a positive drug screen at screening and on retest 1-3 weeks later.
5. The patient had symptoms of mania that may have been attributable to a general medical condition, or secondary to use of medications (eg, corticosteroids)
6. The patient had evidence of any serious and/or unstable neurological illness for which treatment under the auspices of this study would have been contra-indicated.
7. The patient had any serious, unstable medical illness or clinically significant abnormal laboratory assessments that would adversely impact the scientific interpretability or unduly increase the risks of the protocol.
8. The patient had a current general medical condition including neurological disease, diabetes mellitus, thyroid dysfunction, or renal dysfunction that might have been affected adversely by lithium, could have influenced the efficacy or safety of lithium, or would have complicated interpretation of study results.
9. The patient had evidence of current serious homicidal/suicidal ideation such that in the treating physician's opinion it was appropriately safe for the patient to participate in this study.
10. The patient had evidence of current active hallucinations and delusions such that in the treating physician's opinion it was not appropriately safe for the patient to participate in this study.
11. The patient had concomitant prescription of over-the-counter medication or nutritional supplements that would interact with lithium or the patient"s physical or mental status.
12. The patient had any use of psychotropic agents other than stimulants within the preceding 2 weeks, including antipsychotics, monoamine oxidase inhibitors, antidepressants; use of stimulants within the preceding week; or fluoxetine or depot antipsychotics within the past month.
13. The patient had current psychotherapy treatments provided outside the study initiated within 4 weeks prior to screening.
14. The patient had a previous adequate trial with lithium (at least 4 weeks with lithium serum levels between 0.8-1.2 mEq/L).
15. The patient had a history of allergy to lithium.
16. The patient had psychiatric hospitalization within 1 month of screening for psychosis or serious homicidal/serious suicidal ideation.
17. Clinician"s judgment was that the patient was not likely to be able to complete the study as an outpatient due to psychiatric reasons.
18. The patient had a history of lithium intolerance.
19. Females who were currently pregnant or lactating.
20. Sexually active females who, in the investigators" opinion, were not using an adequate form of birth control.
21. Patients who were unable to swallow the study medication.
22. Patients for whom a baseline YMRS score of < 20 was anticipated.
23. Patients with an IQ < 70 (determined using the Wechsler Abbreviated Scales of Intelligence [WASI] Vocabulary and Matrix Reasons Subscales).

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2006-12; Primary Completion 2009-04 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Mean Change in YMRS summary score by treatment | 8 weeks
  Measure of efficacy
Mean change in YMRS parent score | 8 weeks
  Measure of efficacy
Mean change in YMRS child score | 8 weeks
  Measure of efficacy
Rate of treatment emergent adverse events | During administration of study drug
Dosing - PK | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Findling, MD, Principal Investigator — Case Western University
Locations (1):
- CASE Western Reserve University, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Findling RL, McNamara NK, Pavuluri M, Frazier JA, Rynn M, Scheffer R, Kafantaris V, Robb A, DelBello M, Kowatch RA, Rowles BM, Lingler J, Zhao J, Clemons T, Martz K, Anand R, Taylor-Zapata P. Lithium for the Maintenance Treatment of Bipolar I Disorder: A Double-Blind, Placebo-Controlled Discontinuation Study. J Am Acad Child Adolesc Psychiatry. 2019 Feb;58(2):287-296.e4. doi: 10.1016/j.jaac.2018.07.901. Epub 2018 Nov 26. PMID 30738555
- [Derived] Findling RL, Frazier JA, Kafantaris V, Kowatch R, McClellan J, Pavuluri M, Sikich L, Hlastala S, Hooper SR, Demeter CA, Bedoya D, Brownstein B, Taylor-Zapata P. The Collaborative Lithium Trials (CoLT): specific aims, methods, and implementation. Child Adolesc Psychiatry Ment Health. 2008 Aug 12;2(1):21. doi: 10.1186/1753-2000-2-21. PMID 18700004